CLINICAL TRIAL: NCT02552277
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled, Dose Range Finding Study to Access the Efficacy and Safety of Intramuscular Injection of Human Placenta- Derived Cells (PDA-002) in Subjects With Diabetic Peripheral Neuropathy.
Brief Title: A Efficacy and Safety Study of Intramuscular Injection of Human Placenta-Derived Cells (PDA-002) in Subjects With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celularity Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCT-PDA-002-DPN-001
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Nephropathies; Peripheral Nervous System Diseases
Keywords: Diabetic; PDA-002; Placenta-Derived Cells; Peripheral neuropathy; Neuropathy; Double-Blind; Safety; Efficacy; Human Placenta-derived Cells
MeSH Terms: conditions — Diabetic Nephropathies; Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PDA-002 Dose Level 1: 3 x 10^6 cells (Experimental): 3 x 10^6 PDA-002 cells administered intramuscular (IM) on study Days 1, 29, and 57.
  Interventions: Biological: PDA-002
- PDA-002 Dose Level 2: 30 x 10^6 cells (Experimental): 30 x 10^6 PDA-002 cells administered IM on study Days 1, 29, and 57.
  Interventions: Biological: PDA-002
- Placebo (Placebo Comparator): Subjects will receive placebo administered IM on study days 1, 29, and 57.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: PDA-002 — PDA-002 cells administered intramuscular (IM) on study Days 1, 29, and 57.
  Other Names: HUMAN PLACENTA-DERIVED CELLS
  Arms: PDA-002 Dose Level 1: 3 x 10^6 cells; PDA-002 Dose Level 2: 30 x 10^6 cells
Drug: Placebo — Subjects will receive placebo administered on study days 1, 29, and 57.
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, dose range finding study in subjects who have diabetic peripheral neuropathy (DPN). The study will enroll approximately 24 subjects. Subjects will be randomized to receive one of 3 treatments: PDA-002 (3 x 10^6 cells), PDA-002 (30 x 10^6 cells), or placebo (vehicle control) in a 1:1:1 randomization approach. Investigational product or placebo will be administered monthly (3 administrations total on Study Days 1, 29, and 57).

DETAILED DESCRIPTION:
Subjects will undergo a Screening Period (up to 28 days in duration) to determine study eligibility and baseline levels of signs and symptoms of diabetic peripheral neuropathy (DPN) will be established. Subjects will then enter a Treatment Period (6 months in duration). During the Treatment Period, subjects will be evaluated on an ongoing basis (at 8 scheduled study visits). Subjects will receive intramuscular (IM) injections of investigational product (IP) on Study Days 1, 29, and 57 as fifteen 0.30 mL injections (below the knee and above the ankle) in one lower extremity in a blinded manner. After completing the Treatment Period, subjects will enter the Follow-up Period where they will continue to be evaluated at scheduled study visits over the subsequent months.

An analysis of all study data will occur after the last subject has completed Visit 9 (Month 6) and after the last scheduled study visit.

ELIGIBILITY:
Inclusion Criteria: Subjects must satisfy the following criteria to be enrolled in the study:

1. Males and females who are at least 18 years of age at the time of signing the informed consent document.
2. Subject must understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements
4. Diabetes mellitus (DM) Type 2 as defined by the American Diabetes Association (ADA) or World Health Organization (WHO) criteria.
5. Meet established criteria for diabetic peripheral neuropathy (DPN) due to Type 2 diabetes with the following:

   1. Abnormal symptoms 6-item Neuropathy Total Symptom Score (NTSS-6 ≥ 6 points (total score) or ≥ 2.0 points for one or more symptoms) AND
   2. Abnormal signs; Utah Early Neuropathy Scale (UENS) score of 2-24 and/or Neurological Impairment Score of the Lower Limb (NIS-LL) score of 2-10.
6. A female of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to treatment with study therapy. In addition, sexually active Females of Child Bearing Potential (FCBP) must agree to use 2 of the following adequate forms of contraception methods simultaneously such as: oral, inject able, or implantable hormonal contraception, tubal ligation, intrauterine device (IUD), barrier contraceptive with spermicide or vasectomized partner for the duration of the study.
7. Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in sexual activity with FCBP for the duration of the study

Exclusion Criteria: The presence of any of the following will exclude a subject from enrollment:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Other causes of neuropathy in diabetic subjects: chronic inflammatory demyelinating polyneuropathy; neuropathy due to vitamin B12 deficiency, hypothyroidism, and uremia syndrome; and neuropathy due to entrapment or trauma.
3. A reversible course of acute painful diabetic neuropathy syndrome: treatment-induced diabetic neuropathy that presents in the setting of rapid glycemic control; diabetic neuropathic cachexia; and diabetic anorexia, a diabetic neuropathy that is seen with intentional weight loss.
4. History of a prior diagnosis of severe peripheral arterial disease (PAD).
5. Thrombocytopenia and coagulopathy, to avoid severe bruising or bleeding due to multiple intramuscular (IM) injections.
6. Any condition including the presence of laboratory abnormalities that places the subject at unacceptable risk if he or she were to participate in the study.
7. Any condition that confounds the ability to interpret data from the study.
8. Subjects who are taking opioids for the treatment of DPN.
9. Pregnant or lactating females.
10. Subjects with a body mass index > 40 kilgrams (kg)/m^2 at screening.
11. Neuropathy resulting from a condition other than DM and/or significant co-morbid neurological diseases (eg, Parkinson's disease, epilepsy, multiple sclerosis, alcoholic peripheral neuropathy), or exposure to agents suspected to cause symptoms of neuropathy (such as but not limited to metronidazole, antituberculosis medications, and heavy metals).
12. Advanced neuropathy as measured by the absence of sural sensory nerve action potential, or a UENS>24 and or a NIS-LL>10.
13. History of a prior diagnosis of Critical Limb Ischemia.
14. History of diabetic foot ulceration (at any time) and/or or undergoing a limb revascularization procedure(s) and/or amputation(s) due to diabetes mellitus (DM).
15. Diagnosis of Type 1 DM and/or any of the following: diagnosis of DM prior to age 35 years; insulin required to treat DM within 1 year after DM diagnosis; history of diabetic ketoacidosis.
16. Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), or alkaline phosphatase ≥ 2.5 x the upper limit of normal (ULN) at screening.
17. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 at Screening calculated using the Modification of Diet in Renal Disease Study equation or history of an abnormal eGFR < 60 and decline > 15 mL/min/1.73 m2 below normal in the past year.
18. Bilirubin level > 2 mg/dL (unless subject has known Gilbert's disease) at screening.
19. Untreated chronic infection or treatment of any infection with systemic antibiotics within 4 weeks prior to dosing with investigational product (IP).
20. Uncontrolled hypertension (defined as diastolic blood pressure > 100 mmHg or systolic blood pressure > 180 mmHg during screening at 2 independent measurements taken while subject is sitting and resting for at least 5 minutes).
21. History of significant cardiac disorders including but not limited to malignant ventricular arrhythmia, CCS Class III-IV angina pectoris, myocardial infarction/ percutaneous coronary intervention (PCI) / coronary artery bypass graft (CABG) in the 6 months prior to signing the informed consent form (ICF), pending coronary revascularization in the following 3 months, transient ischemic attack/cerebrovascular accident in the 6 months prior to signing the informed consent form, and/or New York Heart Association [NYHA] Stage III or IV congestive heart failure. Note: Stable Canadian Cardiovascular Society (CCS) Class I-II angina is allowed.
22. Poorly controlled DM (hemoglobin A1c > 10%) at screening.
23. Untreated proliferative retinopathy at screening.
24. Life expectancy less than 2 years due to concomitant illnesses.25. History of malignancy within 5 years except for the following circumstances: basal cell or squamous cell carcinoma of the skin, remote history of cancer now considered cured or positive Pap smear with subsequent negative follow-up.

26. History of hypersensitivity to any of the components of the product formulation (including bovine or porcine products, dextran 40, and dimethyl sulfoxide [DMSO]).

27. Subject has received an investigational agent -an agent or device not approved by the US Food and Drug Administration (FDA) for marketed use in any indication- within 90 days (or 5 half-lives, whichever is longer) prior to treatment with study therapy or planned participation in another therapeutic study prior to the completion of this study or has received previous gene or cell therapy at any time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Percent change in the epidermal nerve fiber density (ENFD) at 6 months, compared to baseline | Baseline up to 6 months
  Epidermal nerve fiber density is a measurement used to assess the extent of peripheral diabetic neuropathy. The number of nerve fibers in a skin biopsy will be counted and quantified. A reduction in the number of nerves fibers (EPND)is indicative of worsening neuropathy.

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 2 years
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Koppisetti, Study Director — Celularity Incorporated
Locations (7):
- United States (7):
  - Collaborative Neuroscience Network, LLC- Southland Neurologic Associates - Los Alamitos, Garden Grove, California
  - SDS Clinial Trials, Inc, Orange, California
  - Compass Research, LLC, Orlando, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Nerve And Muscle Center Of Texas, Houston, Texas
  - Endeavor Clinical Trials PA, San Antonio, Texas

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT02552277/Prot_SAP_000.pdf